CLINICAL TRIAL: NCT05879380
Title: MR Pulmonary Angiography to Replace CT Pulmonary Angiography for Patients With a Suspicion of a Pulmonary Embolism
Acronym: MIRACLE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Noordwest Ziekenhuisgroep (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Jos Wallis, Radiologist, Noordwest Ziekenhuisgroep
Other Study IDs: NL90098.029.22
Record Dates: First submitted 2023-04-12; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Embolism; Radiation Exposure
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Suspicion of pulmonary embolism: The group suspected of a pulmonary embolism will receive standard care, consisting of the CTPA to see wether they have a pulmonary embolism or not. Additional to this imaging they will receive a MRPA.
  Interventions: Diagnostic Test: MRPA; Diagnostic Test: CPTA

INTERVENTIONS:
Diagnostic Test: MRPA — patients will receive an extra MRPA, on top of the standard CTPA
Diagnostic Test: CPTA — patients will receive an extra MRPA, on top of the standard CTPA

SUMMARY:
Rational: The first choice of imaging modality for patients with a suspicion of pulmonary embolism is CT pulmonary angiography (CTPA). Our goal is to avoid extra cases of cancer due to the carcinogenic effect of ionizing radiation from using CTPA. This carcinogenic effect is greatest in women under 40. In the Netherlands, at least 100,000 CTPA's are performed each year, 10% of which are in women under 40 years old, resulting in at least 10 extra tumors induced per year. The goal is to investigate whether MR Pulmonary angiography (MRPA) can serve as an alternative to CTPA. If it can replace CTPA, this will result in a significant health benefit.

Objective: the primary objective is to determine the sensitivity and specificity of MR Pulmonary Angiography (MRPA) with CT Pulmonary Angiography (CTPA) as the gold standard.

Secondary outcomes: to determine the clinical applicability of MRPA in daily practice, negative predictive value, positive predictive value, accuracy of MRPA (compared to CTPA), and agreement in assessment between radiologists.

Study design: observational-prospective diagnostic study, an additional MRPA will be performed in patients with a suspicion of pulmonary embolism.

Study population: in patients with clinical suspicion of pulmonary embolism, a standard CTPA is made for exclusion or confirmation of the disease. The study population will consist of 272 patients.

Primary outcome parameters: determining the sensitivity and specificity of MRPA compared to CTPA (gold standard) in patients with a (clinical) suspicion of pulmonary embolism.

Secondary outcome parameters: Determining the negative predictive value, positive predictive value, accuracy, inter-observer agreement with respect to MRPA, and applicability in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent
* 18 years old

Exclusion Criteria:

* Regular exclusion criteria for MR examination,
* Contrast allergy,
* Hemodynamic instability,
* Severe respiratory insufficiency
* Immobile patient.
* Pregnancy
* Dialysis patients
* COVID-19 positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population consists of all patients with a suspicion of pulmonary embolisms on all departments of our hospital - including ER, wards, primary lung-heart aid ward - who undergo a CTPA during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2023-06-02 (Estimated); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | At the end of the study, so probably around February or March 2024. Time frame of approximately 9 months
  To determine the sensitivity of the MRPA towards CTPA, regarding all patients that have been scanned. Then the sensitivity will be calculated and compared to that of the golden standard CTPA
Specificity | At the end of the study, so probably around February or March 2024. Time frame of approximately 9 months
  To determine the specificity of the MRPA towards CTPA. To determine the specificity of the MRPA towards CTPA, regarding all patients that have been scanned. Then the specificity will be calculated and compared to that of the golden standard CTPA

SECONDARY OUTCOMES:
To determine the negative predictive value of MRPA | At the end of the study, so probably around February or March 2024. Time frame of approximately 9 months
  compared to CTPA
To determine the positive predictive value of MRPA | At the end of the study, so probably around February or March 2024. Time frame of approximately 9 months
  compared to CTPA
To determine the accuracy of MRPA | At the end of the study, so probably around February or March 2024. Time frame of approximately 9 months
  compared to CTPA
To determine the inter-observer agreement / variability of MRPA | At the end of the study, so probably around February or March 2024. Time frame of approximately 9 months
  compared to CTPA
To determine the feasibility in daily clinical practice of MRPA | At the end of the study, so probably around February or March 2024. Time frame of approximately 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Remy Geenen, Study Chair — Noordwest Ziekenhuisgroep

IPD SHARING:
Plan to Share IPD: No